CLINICAL TRIAL: NCT05267912
Title: Prospective Multicenter Study Evaluating the Feasibility and Efficacy of Tumor Organoid-based Precision Medicine in Patients With Advanced Refractory Cancers
Brief Title: Prospective Multicenter Study Evaluating Feasibility and Efficacy of Tumor Organoid-based Precision Medicine in Patients With Advanced Refractory Cancers
Acronym: ORGANOTREAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-A00939-32; 2021/3270 (Other: CSET number)
Record Dates: First submitted 2022-02-09; First posted 2022-03-07 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Advanced, Pretreated Solid Tumors
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: * ORGANOTREAT-01: advanced, pretreated colorectal cancer (CRC).
  * ORGANOTREAT-02A: Advanced, pretreated colorectal cancer (CRC) or pancreatic ductal adenocarcinoma (PDAC)
  * ORGANOTREAT-02B: advanced, pretreated solid tumors with a PDO take-on rate ≥50%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ORGANOTREAT 01 (Experimental): To assess the feasibility of timely generating chemograms from PDOs in advanced CRC.
  To assess the proportion of patients treated according to the chemogram tumor board (CTB)'s recommendations on the basis of their personalized chemogram.
  To assess the efficacy and safety of chemogram-driven treatment in advanced CRC.
  Interventions: Procedure: Biopsy
- ORGANOTREAT 02A (Experimental): ORGANOTREAT-02A is a single-arm, Phase II study to evaluate the feasibility of chemogram-driven treatment in patients with advanced, pretreated solid cancers (CRC or PDAC). The primary endpoint is to assess the proportion of patients treated according to the chemogram tumor board (CTB)'s recommendations on the basis of their personalized chemogram.
  Interventions: Procedure: Biopsy
- ORGANOTREAT 02B (Experimental): is a randomized Phase II study to compare the efficacy of chemogram-driven treatment vs SoC in patients with advanced, pretreated solid cancers with a PDO take-on rate ≥50%. A cross-over will allow patients enrolled in the control arm to benefit from chemogram-based treatment. Patients for whom no chemogram can be obtained will not be randomized and they will be treated according to SoC. The primary endpoint will be PFS. The study will include multiple strata, each for a different tumor type (e.g., stratum 1, pancreatic ductal adenocarcinoma (PDAC); stratum 2, CRC; etc.). Each stratum will be conducted and analyzed independently from the other strata.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — We need a biopsy for PDO: PDOs are tridimensional multicellular structures expanded in vitro which retain the genotypic and phenotypic features of their tissue or tumor of origin. PDOs can be exposed to a panel of drugs (chemotherapy, hormonal therapy, targeted therapy) in order to study their sensitivity to each agent (or combination of agents) tested ('chemogram'). Recent studies showed that PDOs can accurately predict the response to treatment of solid tumors and could therefore inform clinical decision on the best therapeutic option for each patient.

SUMMARY:
* PDOs are tridimensional multicellular structures expanded in vitro which retain the genotypic and phenotypic features of their tissue or tumor of origin. PDOs can be exposed to a panel of drugs (chemotherapy, hormonal therapy, targeted therapy) in order to study their sensitivity to each agent (or combination of agents) tested ('chemogram'). Recent studies showed that PDOs can accurately predict the response to treatment of solid tumors and could therefore inform clinical decision on the best therapeutic option for each patient.
* ORGANOTREAT is a multicenter prospective study program of organoid-based precision oncology encompassing 3 studies: ORGANOTREAT-01, a pilot study restricted to advanced CRC, and ORGANOTREAT-02A and -2B, two Phase 2 studies in advanced solid cancers.

DETAILED DESCRIPTION:
ORGANOTREAT-01, -02A and -02B

* Patients with advanced, pretreated solid cancers will be enrolled at the beginning of a standard-of-care (SoC) treatment line to allow sufficient time for PDO (tumor-derived organoid) generation and chemogram.
* A biopsy of an easily accessible tumor site will be performed.
* PDO generation, culture and amplification and drug testing will be performed.
* A chemogram report will be prepared.
* The CTB (Chemogram Tumor Board) will make treatment recommendations based on the chemogram report.
* Patients enrolled in ORGANOTREAT-01, ORGANOTREAT-02A and in the experimental arm of ORGANOTREAT-02B will be treated according to the CTB's recommendations after disease progression or unacceptable toxicity while on SoC.
* Patients will be treated at the investigator's discretion until disease progression or unacceptable toxicities. Patient will be followed until death or study termination, whichever occurs first . Note : Provide, as long as necessary (without time limit) the treatments to patient is agreed by all the centers.
* Patients for whom no chemogram can be obtained will be treated according to Soc

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* ECOG performance status 0-1
* Life expectancy >3 months
* Histologically-confirmed, unresectable, locally advanced or metastatic solid tumor

  * ORGANOTREAT-01: CRC
  * ORGANOTREAT-02A: Colorectal adenocarcinoma (CRC) or pancreatic ductal adenocarcinoma (PDAC)
  * ORGANOTREAT-02B: solid cancers with a PDO take-on rate ≥50%:

    * Stratum 1: PDAC
    * Stratum 2: CRC
    * Other strata: to be added by protocol amendment
* ≥1 measurable lesion according to RECIST v1.1
* ≥1 tumor site accessible to biopsy without significant risk, outside from lung lesion
* Patients are to be biopsied before the start or within the 3 first weeks of the SoC line.
* Failure (disease progression or intolerance) or contraindication to validated treatments in the advanced setting; patients MUST be still eligible for at least 1 (ORGANOTREAT-01 and -2A) or 2 (ORGANOTREAT-02B) validated systemic treatment lines according to approved guidelines:

  * CRC (ORGANOTREAT-01): failure (disease progression or intolerance) or contraindication to fluoropyrimidines, oxaliplatin, irinotecan, anti-EGFR (in RAS wild-type tumors), anti-BRAF (in BRAF V600E mutated tumors), and antiangiogenics; patients must be still eligible for trifluridine-tipiracil and/or regorafenib
  * CRC (ORGANOTREAT-2A): failure (disease progression or intolerance) or contraindication to fluoropyrimidines, oxaliplatin, irinotecan, anti-EGFR (in RAS wild-type tumors), anti-BRAF (in BRAF V600E mutated tumors), and trifluridine-tipiracil/bevacizumab; patients must be still eligible for regorafenib
  * PDAC (ORGANOTREAT-2A): Patients will be included at the beginning of their second line of standard therapy
  * PDAC (ORGANOTREAT-02B stratum 1): patients will be included at the beginning of their first- or second-line of therapy
  * Specifications for supplementary tumor strata in ORGANOTREAT-02 will be defined by protocol amendment
* Adequate hepatic, renal and hematological functions (AST/ALT < 2.5 ULN (5 ULN in cases of liver metastases); Total bilirubin < 1.5 ULN; Albumin > 30 g/L; International normalized ratio (INR) <1.5 ULN; Calculated creatinine clearance >50 mL/min; Absolute neutrophil count >1000/mm3, platelets >100 000/mm3, hemoglobin >9 g/dL) To be performed until 7 days before enrollment
* Informed consent signed by the patient or his/her legal representative
* Affiliation to or beneficiary of a social security system
* A female participant is eligible to participate if she is not pregnant not breastfeeding, and

  1. Not a woman of childbearing potential (WOCBP) OR
  2. A WOCBP should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* A WOCBP must agree to follow the contraceptive guidance or abstain from heterosexual activity during the treatment period and for at least 180 days, after the last dose of treatment.

Exclusion Criteria:

* History of other invasive cancer within 5 years prior to entry into the trial other than adequately treated basal-cell skin cancer or in situ carcinoma of the cervix
* Concomitant medications/comorbidities that may prevent the patient from being biopsied
* Patients with brain or meningeal metastasis, unless definitive therapy occurred more than 6 months ago and with a confirmation of tumoral control and absence of symptoms within 4 weeks of starting study treatment
* Pregnancy or breast-feeding
* Privation of liberty or guardianship
* Geographical, social or psychological reasons precluding study participation and monitoring
* Coagulation abnormality prohibiting a biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2028-01-18 (Estimated); Study Completion 2029-01-18 (Estimated)

PRIMARY OUTCOMES:
ORGANOTREAT-01: Chemogram | 30 months
  number of patients for whom a PDO-based chemogram is obtained within 10 weeks after biopsy
ORGANOTREAT-02A: Proportion of patients treated according to the chemogram tumor board (CTB)'s recommendations on the basis of their personalized chemogram. | 48 months
  Proportion of patients treated according to the chemogram tumor board (CTB)'s recommendations on the basis of their personalized chemogram.
ORGANOTREAT-02B: PFS | 36 months
  progression free survival

SECONDARY OUTCOMES:
ORGANOTREAT-02A and -02B: chemogram | 36 months
  proportion of patients for whom a PDO-based chemogram is obtained within 10 weeks after biopsy,
ORGANOTREAT-01 and -02A: PFS | 36 months
  progression free survival
ORGANOTREAT-01, -02A and -02B: GMI | 36 months
  Growth Modulation Index
ORGANOTREAT-01, -02A and -02B: ORR | 36 months
  Overall Response Rate
ORGANOTREAT-01, -02A and -02B: duration of response | 36 months
ORGANOTREAT-01, -02A and -02B: DCR | 36 months
  Disease Control Rate
ORGANOTREAT-01, -02A and -02B: duration of disease control | 36 months
ORGANOTREAT-01, -02A and -02B: clinical benefit | 36 months
  Clinical benefit (complete response, partial response or stable disease >12 weeks according to RECIST 1.1) in patients treated according to the chemogram results
ORGANOTREAT-01, -02A and -02B: OS | 36 months
  Overall survival
ORGANOTREAT-01, -02A and -02B: Number of chemogram-oriented treatment lines | 36 months
  Number of chemogram-oriented treatment lines

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Jaulin, PhD, Study Director — Gustave Roussy cancer campus
Locations (8):
- France (8):
  - Institut Bergonié, Bordeaux, France
  - Centre Oscar Lambret, Lille, France
  - Centre Léon Bérard, Lyon, France
  - Hôpital Saint Louis, Paris, France
  - Hôpital Pitié-Salpêtrière, Paris, France
  - Institut Godinot, Reims, France
  - Centre Eugène Marquis, Rennes, France
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No